CLINICAL TRIAL: NCT01638338
Title: Optimizing and Integrating the Delivery of Primary Care Services for Risky Drinkers in Region Friuli-Venezia Giulia
Brief Title: Risky Drinkers and the Web: a RCT Study in Region Friuli-Venezia Giulia.
Acronym: EFAR-FVG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Per I Servizi Sanitari N. 2 Isontina (Other)
Collaborators: Ministry of Health, Italy (Other Government); Istituto Superiore di Sanità (Other); University of Leeds (Other); Federsanità, ANCI (Unknown); Codeface Ltd. (Unknown)
Responsible Party: Principal Investigator, Pierluigi Struzzo, MD, MD, Azienda Per I Servizi Sanitari N. 2 Isontina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RF-2010-2318620
Record Dates: First submitted 2012-07-03; First posted 2012-07-11 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Excessive Drinking
Keywords: Alcohol; Risky drinking; Web site; Primary Care; General Practice; Local Community; Mayors
MeSH Terms: interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web site (Experimental): A specific web site for randomization and risky alcohol consumption counseling will be beta tested and created. Risky drinkers allocated to this arm will receive web assisted brief motivational interview.
  They will first be assessed towards risky alcohol consumption and Quality of life (AUDIT and EQ5D). Personal health status will also be assessed with a Likert scale. Brief Intervention will be administered following a consistent number of web pages reporting brief motivational interview Web assisted brief motivational interview on risky drinking
  Interventions: Behavioral: Web assisted brief motivational interview on risky drinking
- Face to Face (Experimental): Risky drinking brief motivational interview provided by the GP.
  Interventions: Behavioral: Face to Face

INTERVENTIONS:
Behavioral: Web assisted brief motivational interview on risky drinking — People allocated to this arm will be given a password to enter and follow a pre-decided set of questions and hints to reduce their drinking
  Other Names: Codeface Ltd.
  Arms: Web site
Behavioral: Face to Face — The counseling provided by the GPs will be done at month 0, 6, 12
  Other Names: Screening and Brief intervention; EIBI; SBI
  Arms: Face to Face

SUMMARY:
The project aims to develop a new approach to risky drinkers by providing a facilitated website access and creating a local integrated support network.

In order to do so:

1) A non inferiority-randomised controlled study will be performed to test the hypothesis that: Brief intervention for risky drinkers delivered in primary care through facilitated access to an alcohol reduction website has non inferior outcomes to face to face brief intervention.

DETAILED DESCRIPTION:
Far from being only an Italian problem, harmful alcohol consumption puts a heavy burden on people's health. Risky behaviors and socio-economical conditions are closely linked and, thus, during critical economical periods, such as this, alcohol related problems increase significantly.

Screening and Brief Intervention is a very effective method to screen and counsel risky people at primary care level but, nevertheless, general practitioners and other health care professionals don't utilize it.

This is mainly due to the fact that the National Health Services should include it into financial agreements for reimbursement or adopt other incentives that, in this critic period, are difficult to be taken into consideration.

What are the alternatives? Utilizing existing resources to propose a different approach at little or no cost: the web and the local communities.

Computers are in almost every house and, if not, the local community can offer their use within libraries or social centres.

Computers are definitely utilized by young people and youngsters are the first to suffer from risky alcohol use. Older people are more and more using them maybe just to surf the web but, if not, its use could be facilitated by their general practitioners.

As stated before, no scientific evidence exists on its effectiveness in respect to the GPs work. For this reason we decided to compare the efficacy of a web based "brief intervention" with a face-to-face brief intervention performed by general practitioners.

We would like to see if a web based approach is, at least, as good as, or not inferior to GPs work.

This project could have an important impact at regional and national level. It could be the starting point of a different way to provide alcohol related health services, utilizing up to date working tools, such as smart phones or iPads, giving a different role to the GPs and improving the action of local social services.

The work of general practitioners could also benefit and more integration with the territorial services could bring to increased visibility of Local Authorities.

The supervision of national and international high-level experts will assure an outstanding quality to the project and the possibility of future inclusion of its results within national or international guidelines for primary care alcohol related services.

This study is a part of a wider community program aiming at involving GPs and Local Authorities for its implementation whose objectives are out of the scope of this RCT.

ELIGIBILITY:
Inclusion Criteria:

* All patients scoring above the agreed cut-point (AUDIT-C: 5 for men and 4 for women) will be invited by their GP to use the trial online consent and assessment module

Exclusion Criteria:

* Patients aged less than 18 years and those who do not give consent will be excluded from the trial and encouraged on-line to make an appointment with their doctor to discuss their drinking habits. Those whose scores indicate dependence will also be excluded from the trial and encouraged on-line to seek additional medical support including referral to a specialist agency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption reduction: Full AUDIT (10 questions) | up to one year
  This measure is referred to the alcohol use reduction

SECONDARY OUTCOMES:
Economic evaluation | one year
  The EQ-5D 5L quality-of-life questionnaire, validated Italian version

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wallace, prof, Study Director — Leeds University; Emanuele Scafato, prof, Study Chair — Istituto Superiore di Sanità
Locations (1):
- Regional Centre for the Training in Primary Care, Monfalcone, Italy

REFERENCES:
- [Derived] Hunter R, Wallace P, Struzzo P, Vedova RD, Scafuri F, Tersar C, Lygidakis C, McGregor R, Scafato E, Freemantle N. Randomised controlled non-inferiority trial of primary care-based facilitated access to an alcohol reduction website: cost-effectiveness analysis. BMJ Open. 2017 Nov 3;7(11):e014577. doi: 10.1136/bmjopen-2016-014577. PMID 29102983
- [Derived] Wallace P, Struzzo P, Della Vedova R, Scafuri F, Tersar C, Lygidakis C, McGregor R, Scafato E, Hunter R, Freemantle N. Randomised controlled non-inferiority trial of primary care-based facilitated access to an alcohol reduction website. BMJ Open. 2017 Nov 3;7(11):e014576. doi: 10.1136/bmjopen-2016-014576. PMID 29102982
- [Derived] Lygidakis C, Wallace P, Tersar C, Marcatto F, Ferrante D, Della Vedova R, Scafuri F, Scafato E, Struzzo P. Download Your Doctor: Implementation of a Digitally Mediated Personal Physician Presence to Enhance Patient Engagement With a Health-Promoting Internet Application. JMIR Res Protoc. 2016 Mar 4;5(1):e36. doi: 10.2196/resprot.5232. PMID 26944482
- See also: Centre for the training in primary care — http://www.ceformed.it